CLINICAL TRIAL: NCT06854068
Title: In-Vivo Evaluation of the Effect of Bioactive Material-Containing Toothpastes and Combined Use of Er-YAG Laser on Dentin Hypersensitivity
Brief Title: Evaluation of the Combined Effect of Bioactive Toothpastes, Desensitizing Agents and Er-YAG Laser on Dentin Hypersensitivity: an In-Vivo Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Principal Investigator, Cem Peskersoy, Doç. Dr., Ege University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E-70198063-050.04-2204953
Record Dates: First submitted 2025-02-25; First posted 2025-03-03 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Dentin Hypersensitivity
Keywords: dentin hypersensitivity; laser; desensitization agent; toothpaste
MeSH Terms: conditions — Dentin Sensitivity | interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: The participants will be aware of which toothpaste they are using; however, they will not know which of their teeth are receiving laser treatment or sensitivity-reducing agents. The evaluator, on the other hand, will be fully informed of all treatments administered.
  The treatment will create the impression that a protective cover is being placed on the other teeth after applying the laser treatment to one tooth, although the laser will only be directed at the specified tooth. Similarly, the sensitivity-reducing agent will be applied to one tooth, while distilled water will be applied to the other sensitive teeth. This approach ensures that the participant will remain unaware of which treatment has been applied to which tooth, allowing for an unbiased assessment of sensitivity.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- G1 Colgate (Active Comparator): Participants with dentin sensitivity in at least three teeth will be divided into four main groups. Subsequently, each of these main groups will be further divided into three subgroups.
  1-) Colgate Sensitivity Pro-Solution (Pro-argin, USA) Subgroup 1a: Laser Subgroup 1b: 3M Clinpro White Varnish (TCP, USA) Subgroup 1c: Control (distilled water)
  Interventions: Device: laser treatment; Device: application of desensitizing agent; Other: Placebo
- G2 Zubio (Active Comparator): 2-) Zubio (Nanohydroxyapatite, Turkey) Subgroup 2a: Laser Subgroup 2b: 3M Clinpro White Varnish (TCP, USA) Subgroup 2c: Control (distilled water)
  Interventions: Device: laser treatment; Device: application of desensitizing agent; Other: Placebo
- G3 Sensodyn (Active Comparator): 3-) Sensodyne Repair and Protect (NovaMin, USA) Subgroup 3a: Laser Subgroup 3b: 3M Clinpro White Varnish (TCP, USA) Subgroup 3c: Control (distilled water)
  Interventions: Device: laser treatment; Device: application of desensitizing agent; Other: Placebo
- G4 GC (Active Comparator): 4-) GC Tooth Mousse (CPP-ACP, Australia) Subgroup 4a: Laser Subgroup 4b: 3M Clinpro White Varnish (TCP, USA) Subgroup 4c: Control (distilled water)
  Interventions: Device: laser treatment; Device: application of desensitizing agent; Other: Placebo

INTERVENTIONS:
Device: laser treatment — In the laser treatment groups, the Fotona LightWalker® Erbium laser (2,940 nm) will be used, with each session lasting five minutes. During treatment, the energy density will be set to 20 J/cm², and the laser tip will be held perpendicular to the target area, applied in continuous and contact modes.
Device: application of desensitizing agent — Mix the product for 15 s. Apply in a thin layer on treatment area(s) with aid of a "microbrush", with no rinsing or removal
Other: Placebo — Simulation of a single layer application (15s) , with the aid of a "microbrush", on the surface of the tooth and with no rinsing or removal.

SUMMARY:
Here's the revised version with the corrected treatment and follow-up session schedule:

---

The aim of this clinical trial is to evaluate the effectiveness of bioactive toothpastes, desensitizing agents, and Er-YAG laser treatments in reducing dentin hypersensitivity. This study also aims to assess the safety and comparative efficiency of these treatment methods. The main research questions are:

* Do bioactive toothpastes, desensitizing agents, and laser treatments individually or in combination reduce dentin hypersensitivity?
* Are there any adverse effects associated with these treatments?

Participants will:

* Be randomly assigned to one of four treatment groups, each using a specific toothpaste (Pro-Argin, Nano-Hydroxyapatite, NovaMin, or CPP-ACP), alongside desensitizing agents, laser treatments, or a placebo.
* Receive two treatment sessions: the first at baseline and the second one week later.
* Attend follow-up evaluations at the 2nd week, 1st month, and 3rd month to assess dentin hypersensitivity using the Visual Analog Scale (VAS) and dental unit air-water sprays.

Researchers will compare the outcomes across groups using statistical analyses (Kolmogorov-Smirnov, Kruskal-Wallis, and Pearson/Spearman tests) to determine the most effective approach for managing dentin hypersensitivity.

DETAILED DESCRIPTION:
In this study, 40 adult patients aged 18 years and older, with at least three teeth affected by dentin hypersensitivity, caries-free, vital, and periodontally healthy, will receive a combination of four different toothpastes, desensitizing agents, and Er-YAG laser treatment. The materials and study groups are organized as follows:

1. **Colgate Sensitive Pro-Relief** (Pro-argin, USA)

   * Subgroup 1a: Laser
   * Subgroup 1b: 3M Clinpro White Varnish (TCP, USA)
   * Subgroup 1c: Control (distilled water)
2. **Zubio** (Nano-hydroxyapatite, Turkey)

   * Subgroup 2a: Laser
   * Subgroup 2b: 3M Clinpro White Varnish (TCP, USA)
   * Subgroup 2c: Control (distilled water)
3. **Sensodyne Repair and Protect** (NovaMin, USA)

   * Subgroup 3a: Laser
   * Subgroup 3b: 3M Clinpro White Varnish (TCP, USA)
   * Subgroup 3c: Control (distilled water)
4. **GC Tooth Mousse** (CPP-ACP, Australia)

   * Subgroup 4a: Laser
   * Subgroup 4b: 3M Clinpro White Varnish (TCP, USA)
   * Subgroup 4c: Control (distilled water)

In the laser treatment groups, the Fotona LightWalker® Erbium laser (2,940 nm) will be used, with each session lasting five minutes. Energy intensity will be set at 20 J/cm², and the laser tip will be positioned perpendicularly to the target area, applied in continuous and contact modes. The desensitizing agent will consist of 3M Clinpro White Varnish containing Tri-Calcium Phosphate (TCP), applied according to the manufacturer's instructions.

Patients who have not used standard fluoride-containing toothpaste for at least one month prior to the study will be excluded to ensure baseline standardization among participants. The assigned toothpaste will be provided to patients according to their group allocation, and they will be instructed to use it three times daily for two minutes each time, without additional oral care products, until their third-month follow-up.

---

Let me know if any additional modifications are needed!

ELIGIBILITY:
Inclusion Criteria:

1. Individuals over the age of 18,
2. Individuals with good oral hygiene,
3. Individuals without systemic contraindications for treatment,
4. Individuals who are reliable for periodic follow-ups, cooperative, and willing to participate in the study,
5. Individuals with sensitivity in at least three teeth,
6. Individuals who have been using a standard toothpaste containing 1100 ppm fluoride for at least one month.

Exclusion Criteria:

1. Individuals with a history of alcohol, drug, or medication addiction,
2. Individuals known to be unable to attend follow-up sessions,
3. Individuals with allergies to any of the products used in the study,
4. Individuals with unstable mental or physical conditions,
5. Pregnant or breastfeeding individuals, as well as those planning pregnancy during the study.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Dentin Hypersensitivity Scores Using VAS at 1 Week, 2 Weeks, 1 Month, and 3 Months After Treatment | Baseline (Pre-treatment), 15 Minutes After Initial Treatment, 1 Week, 2 Weeks, 1 Month, and 3 Months Post-Treatment.
  Reduction in dentin hypersensitivity as assessed by the Visual Analog Scale (VAS) at baseline, immediately after treatment, 1 week, 2 weeks, 1 month, and 3 months post-treatment."

IPD SHARING:
Plan to Share IPD: Yes